CLINICAL TRIAL: NCT03658512
Title: Tübinger Diabetes Mellitus Database (TUEDID)
Status: Recruiting | Type: Observational
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Other Study IDs: 247/2017BO1
Record Dates: First submitted 2018-08-10; First posted 2018-09-05 (Actual); Last update posted 2022-08-29 (Actual); Status verified 2022-08

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- TUEDID cohort

SUMMARY:
Diabetes mellitus is a widespread disease with increasing prevalence worldwide. Patients with diabetes can develop multiple late complications such as neuropathy, retinopathy, nephropathy and cardiovascular comorbidities. So far, there are no reliable predictive tools or markers to estimate if, when and to what extent a patient with diabetes develops late complications. For the patients quality of life and for health economic reasons an improved risk assessment would be desirable. The prospective TUEDID study will characterize diabetic patients to look out for parameters the predict progression of diabetes and its complications.

ELIGIBILITY:
Inclusion Criteria:

* >18 years

Exclusion Criteria:

* no written informed consent

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: People with or without diabetes who are treated at the University Hospital Tübingen
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2018-08-13 (Actual); Primary Completion 2028-02-01 (Estimated); Study Completion 2028-02-01 (Estimated)

PRIMARY OUTCOMES:
Glycemic control (blood glucose) | At enrolment
  Assessed as fasting blood glucose and HbA1C
Glycemic control (HbA1C) | At enrolment
  Assessed as fasting HbA1C

OTHER OUTCOMES:
Liver function | At enrolment
  Parameters for liver function will be assessed (GOT, GPT, AP, Gamma-GT, Lipase, all [U/l])
Renal function | At enrolment
  Parameters for renal function will be assessed (Creatinine, Urea, Cystatin C, all [mg/dl])
Glomerular filtration rate (GFR) | At enrolment
  Glomerular filtration rate will be determined [ml/min/1,73 m²]
Lipid status | At enrolment
  Parameters for evaluation of lipid status will be assessed (LDL, HDL, Cholesterol, triglycerides, all [mg/dl])
Inflammation | At enrolment
  Parameters to evaluate the inflammatory state will be assessed (CRP [mg/dl])
Insulinemia | At enrolment
  Insulin and C-peptide concentrations will be assessed [pmol/l]
Hormones | At enrolment
  Parameters for evaluation of hormonal status will be assessed (TSH [mU/l])
Hormones | At enrolment
  Parameters for evaluation of hormonal status will be assessed (fT3 and fT4 [pmol/l])
Hormones | At enrolment
  Parameters for evaluation of hormonal status will be assessed (Cortisol [nmol/l])
Urine parameters | At enrolment
  Parameters from urine will be assessed (albumin, total protein, both [mg/l])
Urine parameters | At enrolment
  Parameters from urine will be assessed (creatinine [ml/min])
Urine parameters | At enrolment
  Parameters from urine will be assessed (urine sediment via microscopy)
Pancreas | At enrolment
  Lipase and amlyase concentrations for evaluation of pancreas status will be assessed [U/l]
Coagulation | At enrolment
  Parameters for evaluation of coagulation status will be assessed (INR, blood cell count)
Angiological examination | At enrolment
  Angiological examination of parameters for vascular function
Measurement of height and weight | At enrolment
  Height and weight will be measured and reported as BMI (kg/m^2)
Measurement of waist and hip circumference | At enrolment
  Waist and hip circumference will be measured and reported as waist-to-hip ratio
Blood pressure | At enrolment
  Blood pressure will be measured
Heart rate | At enrolment
  Heart rate will be measured
Measurement of advanced glycation endproducts | At enrolment
  Will be assessed by AGE reader
Body composition | At enrolment
  Body fat content and lean mass will be assessed by bioimpedance analysis
Pulmonary function (optional) | At enrolment
  Pulmonary function will optionally be assessed by Spiroergometric Performance Diagnostic
Retinal examination | At enrolment
  Examination of diabetic rethinopathy by fundus photography or optionally by Optical Coherence Tomography Angiography
Anamnestic and Lifestyle questionnaire | At enrolment
  Questions about physical activity, medical history and family background will be asked
cognitive testing | At enrolment
  Cambridge Neuropsychological Test Automated Battery will be performed on tablet
Stool examination (single stool sample) | At enrolment
  composition pof the gut microbiome will be assessed by 16S genome sequencing, bacterial metagenomic analysis, transcriptomics and metabolomics
Macronutrient absorption (optional) | At enrolment
  Stool samples will be collected over multiple days and macronutrient absorption will be assessed by bomb calorimetry
Nasal and skin swab | At enrolment
  nasal and skin swab will be collected and bacterial colonization analysed

CONTACTS AND LOCATIONS:
Locations (1):
- University of Tuebingen, Internal medicine IV, Tübingen, Germany

IPD SHARING:
Plan to Share IPD: No